CLINICAL TRIAL: NCT04534790
Title: Randomized Trial, Anti-inflammatory Effect of Low-Dose Whole-Lung Radiation for COVID-19 Pneumonia
Brief Title: Anti-inflammatory Effect of Low-Dose Whole-Lung Radiation for COVID-19 Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Alejandro Olmos Guzmán, Principal Investigator, MD,, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI-2020-2858
Record Dates: First submitted 2020-08-05; First posted 2020-09-01 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Not radiotherapy (No Intervention): control group
- Radiotherapy (Experimental): patientis with treatment with radiotherapy 1 Gy to Whole lung.
  Interventions: Radiation: Low Dose Radiotherapy

INTERVENTIONS:
Radiation: Low Dose Radiotherapy — anti-inflammatory effect with low-dose radiation to the lungs
  Arms: Radiotherapy

SUMMARY:
There are several clinical studies that mention the benefits of treatment with low-dose radiation therapy to patients with COVID 19, so this study protocol will be started to determine if there is clinical improvement with treatment and low-dose radiation therapy. to all the lung.

DETAILED DESCRIPTION:
Until now, multiple studies with antibiotics and monoclonal antibodies have been used to try to stop this infection, however, the studies have not been conclusive about the real benefit of these drugs, so the search for other alternatives has been an obligation for doctors in all the world. For this reason, it was proposed to carry out a treatment with radiotherapy to the lung based on studies published in the middle of the last century.

In the studies where radiation therapy was given to the lung in cases of infections in the 1930s and 1940s, the most important and with the largest number of patients are the studies by Powel, Scott, Rosseasuy and Openheimer, where together they were treated 594 patients with viral and bacterial infections, obtaining a cure in a total of 524 patients, that is, an 88% chance of cure with this treatment in an average of 7 days.

Treatment with low doses of total lung radiotherapy has not only been used in the treatment of pneumonia in 1930-1940, it has also been used recently in other pathologies such as metaplasia with myeloid myelofibrosis, where they are treated with 1 Gy to both lungs and there is a significant improvement in hypoxia, as well as edema within the first 72 hrs. without presenting side effects due to the treatment at low doses of radiotherapy, control studies were also carried out where it was shown that the low dose of Lung radiotherapy is safe and effective, these studies show that low doses of radiotherapy are safe for patients since it does not generate serious side effects that put the patient's health at risk.

These results are similar to the results obtained in one of the few studies of low-dose total lung radiotherapy in patients with COVID-19, which was performed at Emory University Hospital in Atlanta, where 5 patients with pneumonia, positive for COVID 19 that required supplemental oxygen to which they were given a treatment with radiotherapy 1.5 Gy single dose, at 24 hrs., 4 of the patients rapidly improved clinically, recovering in an average of 1.5 days (range 3 to 96 hrs.). Subsequent imaging and laboratory studies confirmed that low doses of radiation therapy are effective and safe in reducing the symptoms produced by COVID 19.

Recently at the University of Teran in Israel the results of their study were also published, which recruited 5 patients with COVID 19 pneumonia who were oxygen dependent. In this study, a single dose of 0.5 Gy was given, reporting an improvement in 80% of patients and they were discharged from 3 to 7 days.

For which this study was carried out with the objective of determine the anti-inflammatory effect of low-dose total lung radiation therapy in patients with respiratory distress syndrome secondary to covid-19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes
2. Age > 18 years
3. Laboratory confirmation of SARS-CoV-2 infection
4. Acute Respiratory Distress Syndrome in any degree with a hospital treatment requirement.

Exclusion Criteria:

1. Patients who do not agree to receive the treatment
2. Sepsis data
3. Hemodynamic instability

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | 7 days
  improvement of oxygen saturation

SECONDARY OUTCOMES:
improvement of laboratory and imaging parameters | 7 -14 days
  improvement in acute phase reactants and simple tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Social Secure Mexican Institute, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Undecided